CLINICAL TRIAL: NCT00109525
Title: Early Diagnosis of Nosocomial Candidiasis Study
Brief Title: Early Diagnosis of Candidiasis in Premature Infants
Acronym: Candida
Status: Completed | Type: Observational
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Center for Research Resources (NCRR) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: NICHD-NRN-0030; UL1RR024139 (NIH); UL1RR024160 (NIH); M01RR016587 (NIH); M01RR000030 (NIH); M01RR000032 (NIH); M01RR000039 (NIH); M01RR000044 (NIH); M01RR000054 (NIH); M01RR000059 (NIH); M01RR006022 (NIH); M01RR000633 (NIH); M01RR000070 (NIH); M01RR007122 (NIH); M01RR000750 (NIH); M01RR000080 (NIH); M01RR008084 (NIH); M01RR000997 (NIH); U10HD036790 (NIH); U10HD021364 (NIH); U10HD021373 (NIH); U10HD021385 (NIH); U10HD021397 (NIH); U10HD027851 (NIH); U10HD027853 (NIH); U10HD027856 (NIH); U10HD027871 (NIH); U10HD027880 (NIH); U10HD027904 (NIH); U10HD034216 (NIH); U10HD040461 (NIH); U10HD040492 (NIH); U10HD040498 (NIH); U10HD040521 (NIH); U10HD040689 (NIH); U10HD053089 (NIH); U10HD053109 (NIH); U10HD053119 (NIH)
Record Dates: First submitted 2005-04-28; First posted 2005-04-29 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Infection; Candida; Candidiasis; Infant, Newborn; Infant, Low Birth Weight; Infant, Small for Gestational Age; Infant, Premature
Keywords: NICHD Neonatal Research Network; Fungal Infection; Mycosis; Extremely Low Birth Weight (ELBW); Prematurity; Clinical Judgement; Polymerase chain reaction (PCR) testing; Beta-glucan assay; Mass Spectrometry; Lumbar puncture
MeSH Terms: conditions — Infections; Torulopsis; Candidiasis; Premature Birth; Mycoses; Pathologic Complete Response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This observational study evaluated the performance of new lab tests in detecting candida species fungal infections in extremely low birth weight (ELBW) infants quickly and accurately. 19 NICHD Neonatal Research Network sites enrolled 1,500 infants with birth weights ≤1,000g; 100 of these infants later tested positive for candidiasis. Blood, urine, and lumbar puncture samples were collected whenever other specimens were obtained from participants for cultures. These samples are being tested using the new methods and compared with standard culture results. Surviving study subjects completed a neurodevelopmental evaluation at 18-22 months corrected age.

DETAILED DESCRIPTION:
Candida species are a leading cause of infectious mortality in newborns with the incidence rates estimated at 4-18% in extremely low birth weight (ELBW) infants. 20-30% of these infants are likely to die. Because candida can invade virtually all body tissues (eyes, brain, heart, lung, liver, spleen, urinary tract, and joints), survivors of invasive Candida infections are at risk of blindness, developmental delays, and the need for surgical and other corrective procedures.

Time is of the essence in detecting and treating these infections, with infant mortality from candidiasis largely attributed to duration of time for cultures to become positive for Candida. Diagnosis of candidiasis is challenging - blood and urine tests are slow (taking up to 72 hours to complete) and inaccurate in many cases, showing negative results despite overwhelming disease in adults as well as children. These problems are likely made worse in neonates, with smaller amounts of blood available for testing and infections that often spread to tissues inaccessible for testing.

This observational study is evaluating the performance of new lab tests (beta-glucan assays, Gas Chromatography Mass Spectrometry for D-arabinitol, and polymerase chain reaction tests) compared to existing culture tests in detecting candida species fungal infections in extremely low birth weight (ELBW) infants quickly and accurately.

In this study, 19 NICHD Neonatal Research Network sites enrolled 1,500 infants with birth weights ≤1,000g by 72 hours of life; more than 100 of these infants later tested positive for candidiasis. In the larger cohort, whenever cultures of blood or urine were obtained, or a lumbar puncture was done, additional samples and clinical data were collected. These additional samples are being tested using the new techniques under investigation. No additional blood specimens were taken once participants had a positive blood culture for candida. Note: Test procedure reagents are being provided the Duke University laboratory by Cape Cod Incorporated and Rockeby; the Thrasher Research Fund is also providing support to the Duke University laboratory.

Surviving study subjects completed a neurodevelopmental evaluation at 18-22 months corrected age to evaluate potential early risk factors with long-term outcome.

ELIGIBILITY:
Inclusion Criteria:

* Infants born ≤1,000g birth weight
* Infants >72 hours old and less than 120 days old

Exclusion Criteria:

* Prior positive blood culture for Candida
* Evidence of congenital candidiasis
* Parents/legal guardians refuse consent

Ages: 3 Days to 120 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants with birth weights ≤1,000 grams
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2004-03; Primary Completion 2007-07 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Probability of invasive candidiasis based on new assay results | Until discharge
Determine test performance of clinical predictive model | Until discharge

SECONDARY OUTCOMES:
Determine test performance (sensitivity and specificity) of polymerase chain reaction (PCR) testing | Until discharge
Determine test performance of Beta-glucan assay | Until discharge
Determine test performance of Gas Chromatography Mass Spectrometry for D-arabinitol of blood samples | Until discharge
Determine test performance of Gas Chromatography Mass Spectrometry for D-arabinitol of urine samples | Until discharge
Determine test performance of the blood culture | Until discharge
Determine test performance of the lumbar puncture (cell count, protein, glucose, and culture) | Until discharge
Determine test performance of tracheal aspirates | Until discharge
Determine test performance of urine cultures | Until discharge
Compare clinical predictive model performance to neonatologist clinical judgment | Until discharge
Determine incidence of end-organ damage in neonates with candidemia | Until discharge
Determine resistance patterns of organisms isolated | Until discharge
Determine molecular epidemiology of candidemia | Until discharge
Determine genetic expression of organism virulence factors | Until discharge
Neurodevelopmental outcome | 18-22 months corrected age

CONTACTS AND LOCATIONS:
Overall Officials: Abbot R. Laptook, MD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; Michele C. Walsh, MD MS, Principal Investigator — Case Western Reserve University, Rainbow Babies and Children's Hospital; Ronald N. Goldberg, MD, Principal Investigator — Duke University; Barbara J. Stoll, MD, Principal Investigator — Emory University; Brenda B. Poindexter, MD MS, Principal Investigator — Indiana University; Abhik Das, PhD, Principal Investigator — RTI International; Krisa P. Van Meurs, MD, Principal Investigator — Stanford University; Ivan D. Frantz III, MD, Principal Investigator — Tufts Medical Center; Waldemar A. Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Neil N. Finer, MD, Principal Investigator — University of California, San Diego; Kurt Schibler, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Edward F. Bell, MD, Principal Investigator — University of Iowa; Shahnaz Duara, MD, Principal Investigator — University of Miami; Kristi L. Watterberg, MD, Principal Investigator — University of New Mexico; Dale L. Phelps, MD, Principal Investigator — University of Rochester; Kathleen A. Kennedy, MD MPH, Principal Investigator — The University of Texas Health Science Center, Houston; Pablo J. Sanchez, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas; T. Michael O'Shea, MD MPH, Principal Investigator — Wake Forest University; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Richard A. Ehrenkranz, MD, Principal Investigator — Yale University
Locations (20):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - University of California at San Diego, San Diego, California
  - Yale University, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Tufts Medical Center, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - Wake Forest University, Charlotte, North Carolina
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas

REFERENCES:
- [Result] Benjamin DK Jr, Stoll BJ, Gantz MG, Walsh MC, Sanchez PJ, Das A, Shankaran S, Higgins RD, Auten KJ, Miller NA, Walsh TJ, Laptook AR, Carlo WA, Kennedy KA, Finer NN, Duara S, Schibler K, Chapman RL, Van Meurs KP, Frantz ID 3rd, Phelps DL, Poindexter BB, Bell EF, O'Shea TM, Watterberg KL, Goldberg RN; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Neonatal candidiasis: epidemiology, risk factors, and clinical judgment. Pediatrics. 2010 Oct;126(4):e865-73. doi: 10.1542/peds.2009-3412. Epub 2010 Sep 27. PMID 20876174
- [Result] Adams-Chapman I, Bann CM, Das A, Goldberg RN, Stoll BJ, Walsh MC, Sanchez PJ, Higgins RD, Shankaran S, Watterberg KL, Duara S, Miller NA, Heyne RJ, Peralta-Carcelen M, Goldstein RF, Steichen JJ, Bauer CR, Hintz SR, Evans PW, Acarregui MJ, Myers GJ, Vohr BR, Wilson-Costello DE, Pappas A, Vaucher YE, Ehrenkranz RA, McGowan EC, Dillard RG, Fuller J, Benjamin DK Jr; Eunice Kennedy Shriver National Institutes of Child Health and Human Development Neonatal Research Network. Neurodevelopmental outcome of extremely low birth weight infants with Candida infection. J Pediatr. 2013 Oct;163(4):961-7.e3. doi: 10.1016/j.jpeds.2013.04.034. Epub 2013 May 30. PMID 23726546
- [Result] Bliss JM, Wong AY, Bhak G, Laforce-Nesbitt SS, Taylor S, Tan S, Stoll BJ, Higgins RD, Shankaran S, Benjamin DK Jr; Candida Subcommittee of the Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Candida virulence properties and adverse clinical outcomes in neonatal candidiasis. J Pediatr. 2012 Sep;161(3):441-447.e2. doi: 10.1016/j.jpeds.2012.02.051. Epub 2012 Apr 14. PMID 22504098
- [Result] Greenberg RG, Benjamin DK Jr, Gantz MG, Cotten CM, Stoll BJ, Walsh MC, Sanchez PJ, Shankaran S, Das A, Higgins RD, Miller NA, Auten KJ, Walsh TJ, Laptook AR, Carlo WA, Kennedy KA, Finer NN, Duara S, Schibler K, Ehrenkranz RA, Van Meurs KP, Frantz ID 3rd, Phelps DL, Poindexter BB, Bell EF, O'Shea TM, Watterberg KL, Goldberg RN, Smith PB; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Empiric antifungal therapy and outcomes in extremely low birth weight infants with invasive candidiasis. J Pediatr. 2012 Aug;161(2):264-9.e2. doi: 10.1016/j.jpeds.2012.01.053. Epub 2012 Mar 15. PMID 22424952
- [Result] Wynn JL, Tan S, Gantz MG, Das A, Goldberg RN, Adams-Chapman I, Stoll BJ, Shankaran S, Walsh MC, Auten KJ, Miller NA, Sanchez PJ, Higgins RD, Cotten CM, Smith PB, Benjamin DK Jr; NICHD Neonatal Research Network. Outcomes following candiduria in extremely low birth weight infants. Clin Infect Dis. 2012 Feb 1;54(3):331-9. doi: 10.1093/cid/cir800. Epub 2011 Dec 5. PMID 22144537
- See also: NICHD Neonatal Research Network — https://neonatal.rti.org/